CLINICAL TRIAL: NCT03482505
Title: Rainbow Acoustic Monitoring (RAM) in Patients Weighing up to 10kg Comparison Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SZMU0011
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Respiration Rate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- INVSENSOR00004 (Experimental): All enrolled subjects will receive the INVSENSOR00004 sensor. The INVSENSOR00004 rainbow acoustic monitoring (RAM) acoustic respiration sensor is designed to noninvasively convert acoustical airflow patterns into respiratory rate (RRa).
  Interventions: Device: INVSENSOR00004

INTERVENTIONS:
Device: INVSENSOR00004 — The INVSENSOR00004 will be placed on the subject's neck or chest to provide acoustic respiration rate.

SUMMARY:
The objective of this clinical investigational study is to compare the acoustic respiration rates (RRa) obtained using the INVSENSOR0004 sensor in the subjects up to 10 kg with the respiration rates determined by manual annotations (RRref), and when applicable with capnography respiration rate (RRcap).

ELIGIBILITY:
Inclusion Criteria:

* Subjects weighing up to 10kg
* Subjects will be inpatients and/or outpatients admitted to the NICU (Neonatal Intensive Care Unit) or PICU (Pediatric Intensive Care Unit) or PACU (Post-Anaesthesia Care Unit)
* The parent/legal guardian has given written informed consent/assent to participate in the study.

Exclusion Criteria:

* Subjects with underdeveloped skin
* Subjects with skin abnormalities at the planned application sites that may interfere with sensor application, per directions-for-use (DFU) or trans-illumination of the site, such as burns, scar tissue, infections, abnormalities, etc.
* Subjects deemed not suitable for the study at the discretion of the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Medical Center Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00004
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00004
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Acoustic Respiration Rate (RRa)
Description: Acoustic respiration rate (RRa) as determined by the INVSENSOR00004 will be compared to measurements of actual respiration rates as determined by manual annotation of recorded respiration waveform (RRref) data. Evaluation of the RRa measurements will be reported as bias between the RRa and the RRref.
Time Frame: One study visit lasting up to 60 minutes.
Population: Sufficient number of cases to meet sample size criteria for assessing outcomes was not achieved. The protocol required a minimum of 18 subjects with valid breaths to calculate the bias, precision, and ARMS of the study. This study was not able to meet this target and therefore the bias, precision, and ARMS could not be calculated (primary outcome measure).
Arm/Group | INVSENSOR00004
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 60 minutes.
Arm/Group | INVSENSOR00004
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT03482505/Prot_SAP_000.pdf